CLINICAL TRIAL: NCT05454189
Title: A Prospective, Randomized Study To Evaluate The Safety of Extending The Routine Flushing Of Implanted Port Devices From 4 Weeks To 12 Weeks
Brief Title: Safety of Extending The Routine Flushing Of Implanted Port Devices From 4 Weeks To 12
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essentia Health (Other)
Collaborators: Minnesota Cancer Clinical Trials Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MNCCTN024; EH21C1 (Other: Essentia Health); EH22738 (Other: Essentia Health)
Record Dates: First submitted 2022-06-24; First posted 2022-07-12 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Maintenance of Implanted Port Devices

STUDY DESIGN:
Intervention Model Description: The study is a prospective, randomized study to determine the non-inferiority of every 12 week IPD flushes compared to every 4 week flushes in participants on an IPD maintenance flush schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 4-week IPD Flushing Schedule (Active Comparator): IPD standard maintenance flushes and port assessments every 4 weeks.
  Interventions: Device: Standard IPD Flush Schedule
- 12-week IPD Flushing Schedule (Experimental): IPD standard maintenance flushes and port assessments every 12 weeks.
  Interventions: Device: Reduced IPD Flush Schedule

INTERVENTIONS:
Device: Reduced IPD Flush Schedule — IPD flush every 12 weeks
  Arms: 12-week IPD Flushing Schedule
Device: Standard IPD Flush Schedule — IPD flush every 4 weeks
  Arms: 4-week IPD Flushing Schedule

SUMMARY:
Implanted port devices (IPD) play an essential role in the safe administration of cancer treatments by providing a device to safely administer caustic chemotherapy agents. The current recommended frequency of flushing the IPD per manufacturers guidelines is every 4-6 weeks. The purpose of this study is to find out if extending IPD flushes to every 12 weeks is safe and if it is just as effective as every 4 week flushing.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving written informed consent will complete port specific histories, assessments and questionnaires within 14 days prior to registration. Eligible, consented participants will be registered to the study and randomized to receive either IPD standard maintenance flushes and port assessments every 4 weeks or every 12 weeks for an initial 12 week interval. If study participants agree to the continuation portion of the study, they will continue to receive either IPD standard maintenance flushes and port assessments every 4 weeks or every 12 weeks for up to an additional three 12 week cycles.

ELIGIBILITY:
Inclusion Criteria:

* Hematology/Oncology patients ≥ 18 years old with an Implanted Port Device.
* No planned clinical visits for at least 12 weeks.
* No planned need to access Implanted Port Device within next 12 weeks outside of routine flushing. Potential reasons to access can include but are not limited to lab draw, infusion, IV contrast.
* No planned removal of IPD within 12 weeks of registration.
* No Deep Vein Thrombosis or significant Implanted Port Device complication within ≤ 4 weeks of registration.
* Patient Implanted Port Device with documented blood return ≤ 14 days of registration.
* Ability to read and speak English.
* Able to give informed consent.

Exclusion Criteria:

* Allergy to heparin
* Vulnerable populations: pregnant women, prisoners, mentally handicapped.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of IPD patency | 12 weeks post randomization
  IPD patency without major complication

SECONDARY OUTCOMES:
Long-term rate of IPD patency in scheduled 4-week versus 12-week IPD flushes at 24,36 and 48 weeks post randomization. | Up to 48 weeks post randomization
  Rate of IPD patency during long term follow-up
Difference in complication rates in scheduled 4-week versus 12-week IPD flushes at 12, 24,36 and 48 weeks post randomization. | Up to 48 weeks post randomization
  Differences in specific complications such as occlusion, infection, mechanical as assessed by port assessments and adverse events
Difference in healthcare and patient cost in scheduled 4-week versus 12-week IPD flushes | Up to 48 weeks post randomization
  Determine healthcare and patient cost differences based documented participant charges and participant reported responses to a 8 question financial burden questionnaire. The questionnaire gathers demographic information about employment, method of payment, estimated costs, education level, and smoking status.
Change in Participant Quality of Life and Satisfaction in Scheduled 4-week versus 12 week IPD flushes | Up to 48 weeks post randomization
  Compare participant quality of life and satisfaction over time and between 4-week versus 12-week IPD flushes as assessed by participant responses to 7 question quality of life questionnaire. The questionnaire is specific to IPD flushing and uses a 5 point likert scale.
Impact of smoking, participant age, IPD age, and concomitant medications on complication rates in scheduled 4-week versus 12 week IPD flushes. | Up to 48 weeks post randomization
  Impact of smoking, participant age, IPD age, and concomitant medications on complication rates as assessed by participant response smoking status and port assessments and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bret Friday, MD, PhD, Principal Investigator — Essentia Health
Locations (17):
- United States (17):
  - Mayo Clinic Health System - Albert Lea, Albert Lea, Minnesota
  - Essentia Health St. Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health Deer River Clinic, Deer River, Minnesota
  - Essentia Health St Mary's Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Duluth Clinic, Duluth, Minnesota
  - Essentia Health Fosston, Fosston, Minnesota
  - Fairview Grand Itasca Clinic & Hospital, Grand Rapids, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Range Medical Center, Hibbing, Minnesota
  - Mayo Clinic Health System - Mankato, Mankato, Minnesota
  - Monticello Cancer center, Monticello, Minnesota
  - Essentia Health Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Sanford Worthington Medical Center, Worthington, Minnesota
  - Essentia Health Fargo, Fargo, North Dakota

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical plan and consent form will be available on request. Data will be available on aggregate level; data will be deidentified, the full dataset and statistical code will be available upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after study completion and for 36 months
Access Criteria: A full description of the intended use of the data must be sent to the Project Direct for review and approval. Participant consent for data sharing is conditioned and new ethics approval may be required.